CLINICAL TRIAL: NCT07071038
Title: The 'SWIVEL' Study (Switch Vs Effects Relief): Effectiveness of a Medication 'Switch' vs Guideline-Directed Interventions for Relieving Side Effects of Aromatase Inhibitors Among Breast Cancer Patients
Brief Title: Evaluating the Use of a Medication 'Switch' vs Guideline-directed Interventions for Relieving Side Effects of Aromatase Inhibitors Among Breast Cancer Patients
Acronym: SWIVEL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Elaine.P.Kuhn, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Study02001994; 23KUH994 (Other: Dartmouth Cancer Center, Dartmouth Hitchcock); NCI-2025-09080 (Other: NCI ID)
Record Dates: First submitted 2025-06-23; First posted 2025-07-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Adjuvant Treatment; Early Stage Breast Cancer
Keywords: breast cancer surgery; aromatase inhibitor; aromatase side effects; hormone therapy; quality of life; adherence; early breast cancer; switching medications; hormonal therapy; letrozole; anastrozole; exemestane; tamoxifen; adjuvant therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is phase II, randomized-controlled trial with option for cross-over that compares the effectiveness of a 'switch' in hormonal therapy to guideline-directed intervention (GDI) for frontline management of side effects of aromatase inhibitors among breast cancer patients. After starting AI, participants will be contacted at 2 weeks, and then every 4-weeks to screen for development of bothersome side effects using a validated screening tool. Participants with a positive screen will receive standard of care advice for managing side effects, and in addition will be randomized 1:1 to either receiving a different AI ("switch") or GDI. In addition to baseline, surveys will be administered at time of positive screening (randomization), and 3- and 6-months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Switch (Active Comparator): Participants (people taking part in this study) enrolled to this study will receive treatment with the aromatase inhibitor (AI) Letrozole and fill out surveys to check for side effects to see how the side effects are making their daily life harder. If side effects are reported, the Participant will be randomized (placed by chance) to a group where they will receive either a different AI ('switch') or receive guideline directed intervention "GDI" using medication and non-medication treatment options.
  Interventions: Drug: Switch
- Guideline Directed Intervention (GDI) (Active Comparator): Participants will receive evidence-based (proven to work) treatment options for side effects according to national guidelines; these may include medications or non-medication options (guideline-directed interventions, GDIs).
  Interventions: Other: Guideline Directed Intervention (GDI)

INTERVENTIONS:
Drug: Switch — Participants in the switch arm will receive a new prescription for either anastrozole or exemestane at a dose of 1mg or 25mg daily, respectively. The choice of AI in the first line setting will be at the discretion of the treating oncologist. If side effects persist after the 1st line switch, the participant will have the option to switch to another AI not yet tried, or to tamoxifen at 20mg daily
  Arms: Switch
Other: Guideline Directed Intervention (GDI) — Subjects in this group will receive a guideline-directed intervention "GDI" using medication and/or non-medication treatment options according to the National Comprehensive Cancer Network (NCCN) supportive care guidelines. A GDI Book was created for this trial that lists treatment options and resources for each of the common side effects of hormonal therapy and is available for providers and staff to help select treatment options. For less common side effects with limited evidence-based options, treatment will be determined in collaboration with the treating provider and PI, using best available evidence.
  Arms: Guideline Directed Intervention (GDI)

SUMMARY:
Researchers have learned that about 50% of women do not finish the standard 5-year breast cancer treatment with an aromatase inhibitor. An aromatase inhibitor is hormone therapy that lowers the chance of breast cancer coming back (recurring) after surgery by blocking an enzyme in fat tissue called aromatase; aromatase changes other hormones in the body to estrogen. Women who do not complete the standard 5-year treatment are at higher risk of their cancer coming back. The goal of this research is to prevent breast cancer from coming back after surgery by helping women to stay on treatment with aromatase inhibitors. Researchers believe the best path to help women to stay on treatment is to create a better way to manage (control) side effects.

DETAILED DESCRIPTION:
This is a two-arm, randomized-controlled trial with option for cross-over that compares the effectiveness of a 'switch' in hormonal therapy to guideline-directed intervention (GDI) for frontline management of side effects of aromatase inhibitors among breast cancer patients. Researchers plan to enroll post-menopausal patients with breast cancer who receive a first-time prescription for an aromatase inhibitor (AI). The anticipated enrollment is 124 participants to meet the goal of 62 evaluable participants.

Baseline symptom burden and quality of life will be assessed by validated surveys prior to starting AI. After starting AI, participants will be contacted at 2 weeks, and then every 4-weeks to screen for the development of bothersome side effects using a validated screening tool. The screening tool (FACIT GP5) is a single-item questionnaire that asks participants to respond to the following: "I am bothered by side effects of treatment," with answers ranging from 'Not at all' (score 0) to 'Very much' (score 4). Participants who score either a 3 or 4 on the FACIT GP5 will be considered to have a positive screening result. They will be randomized 1:1 to either receiving a different AI ('switch') or guideline-directed intervention (GDI). A 'GDI Book' was created for this study and will serve as a reference for selecting GDI treatment.

Participants who continue to have symptoms despite completing two lines of treatment within their assigned arm will be allowed to cross-over to the other treatment arm. Patients who are otherwise doing well in their treatment arm may stay in that treatment arm for the duration of the study. Cross-over is entirely optional.

Participants who do not develop side effects will continue to be monitored on study for up to 6 months. Participants with side effects that do not meet criteria for randomization (FACIT GP5 scores of 1 or 2) will receive standard of care at the discretion their treating provider.

Urine samples will be collected as a part of this study, to assess for adherence to endocrine therapy at the time of randomization, and at 3, 6 12 and 24 months after randomization. For participants that are not randomized, urine will be collected at 6, 12 and 24 months only. Urine samples will be collected during routine office visits when possible. Urine test results will remain anonymous (the treating provider will not know the results).

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of DCIS or invasive breast cancer by core needle or incisional biopsy.
* The DCIS or invasive cancer must be estrogen receptor alpha (ER)-positive
* The invasive cancer must be HER2-negative (IHC 0-1+, or with a FISH ratio of <1.8 if IHC is 2+ or if IHC has not been done)
* Clinical Stage I-III invasive breast cancer or DCIS
* Patients for whom adjuvant treatment with one of the following would be clinically indicated: letrozole, anastrozole, exemestane
* Patients who anticipate continuing with adjuvant endocrine therapy for a minimum of 2 years at the time of registration
* Women over 18 years of age who are post-menopausal, defined as last menstrual period >2 years prior to registration, or >1 year prior to registration with FSH and estradiol in post-menopausal range.
* Patients must meet the following clinical laboratory criteria:

  * Absolute neutrophil count (ANC) >1,000/mm3 and platelet count > 75,000/mm3
  * Total bilirubin <1.5 x the upper limit of the normal range (ULN).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN.
* Ability to give informed consent.

Exclusion Criteria:

* Prior endocrine therapy for any histologically-confirmed cancer or prevention of breast cancer in the last 10 years is not allowed.
* Any other adjuvant therapy for breast cancer. Exception: Bisphosphonate or denosumab treatment for metabolic bone issues are allowed.
* Patients who are prescribed tamoxifen as the first endocrine therapy rather than an aromatase inhibitor.
* Women who are pregnant or lactating.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2027-08-05 (Estimated)

PRIMARY OUTCOMES:
Change in Endocrine Symptom Burden at 3 months | 3 months after randomization
  The primary outcome of this study is the change in the Functional Assessment of Cancer Therapy Endocrine Subscale (FACT-ES) endocrine symptom subscale (ESS-23) survey score as measured from the time of randomization to 3 months, or at the time of cross-over or discontinuation of AI due to intolerable side effects, whichever comes first. The ESS-23 score ranges from 0-92, with lower scores indicating higher symptom burden.

SECONDARY OUTCOMES:
Change in Symptom Burden at 3 and 6 months (FACT-ES) | 3 and 6 months after randomization
  Change in FACT-ES Endocrine Subscale survey scores from time to randomization to 3-months and at 6 months, after allowing for cross-over in an intention to treat analysis
Change in Symptom Burden at 3 and 6 months (PROMIS) | 3 and 6 months
  Change in Patient-Reported Outcomes Measurement Information System (PROMIS) survey scores (fatigue, depression, anxiety, pain, sleep disturbance, physical function) from baseline to 3 and 6 months in an intention to treat analysis. Each PROMIS short form symptom survey consists of 8 items, and raw scores are converted to T-scores ranging from 0-100 with associated standard errors based on the general US population. Higher T scores correspond to more symptom burden. The change in average T scores for relevant symptom surveys will be compared between groups.
Change in Symptom Burden at 3 and 6 Months (FSFI) | 3 and 6 months
  Change in Female Sexual Function Index (FSFI) survey score from baseline to 3 and 6 months in an intention to treat analysis. The FSFI is a 19-item validated survey, answers are given on a 5-point Likert scale and questions are weighted to give a total score ranging from 2-36, with higher scores indicating better sexual function.
Quality of life at 3 and 6 months | 3 and 6 months after randomization
  Change in the Functional Assessment of Cancer Therapy-General (FACT-G) survey score from time to randomization to 3- and 6-months. The FACT-G measures physical, social, emotional and function well-being, with a total of 27 items that are answered on a 5-point Likert scale. Total scores range from 0-108, with higher scores indicating better quality of life.
Adherence to Endocrine Therapy at 3 and 6 months | 3 and 6 months after randomization
  Adherence to endocrine therapy will be assessed by urine testing and corroborated by VOILS survey and pharmacy records. The VOILS Adherence scale assesses patient-reported extent and reasons for nonadherence. Answers are given on a 5-point Likert scale, with higher scores indicating a greater degree of non-adherence.
Long-Term Adherence to Endocrine Therapy at 12 and 24 months | 12 and 24 months after randomization
  Long-term adherence to endocrine therapy will be assessed by urine testing and corroborated by VOILS survey and pharmacy records.
Factors Associated with Adherence to Endocrine Therapy | 2 years after randomization
  Patient-perceived self-efficacy, illness perception and hopefulness will be evaluated using validated surveys at the time of enrollment. Those survey scores will be assessed for associations with long-term adherence to endocrine therapy.
Distant Disease-Free Survival at 1, 2 and 5 Years | 5 years after randomization
  Distant disease-free survival will be assessed by chart review at 1, 2, and 5 years after randomization.

OTHER OUTCOMES:
TSQM Screening Tool | 2 years after enrollment
  A modified version of the Treatment Satisfaction Questionnaire for Medication (TSQM) will be assessed as a screening tool to identify patients who are having clinically meaningful side effects requiring intervention.
Responder Thresholds to Define Clinically Meaningful Change in Symptoms | 3 and 6 months after randomization
  Symptom surveys have classically been assessed over time using the 'minimally important difference' (MID) to define clinically meaningful results. This exploratory objective will test the sensitivity of a predefined 'responder threshold' (score change) to identify participants with clinically meaningful improvement in symptoms, according to recent FDA recommendations.
Disparities and Access to Care | 6 months after randomization
  Patient perceived barriers to the use of evidence-based interventions will be assessed by exit survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided